CLINICAL TRIAL: NCT05210686
Title: Clinical and Biochemical Effects of the Adjunctive Use of a Polynucleotides and Hyaluronic Acid Based Gel in the Subgingival Re-instrumentation of Residual Periodontal Pockets: a Randomized, Split-mouth Clinical Trial.
Brief Title: Effects of Polynucleotides and Hyaluronic Acid Based Subgingival Periodontal Pockets Re-instrumentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Chairman Section of Periodontics Director of Master Program in Periodontics, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 4766 Prot n 947/17
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Periodontal Pocket
MeSH Terms: conditions — Periodontal Pocket

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- subgingival re-instrumentation + gel containing PDRN and HA (Experimental): subgingival re-instrumentation + gel containing PDRN and HA
  Interventions: Other: subgingival re-instrumentation
- subgingival re-instrumentation (Active Comparator): subgingival re-instrumentation
  Interventions: Other: subgingival re-instrumentation

INTERVENTIONS:
Other: subgingival re-instrumentation — subgingival re-instrumentation (control)

SUMMARY:
The purpose of this randomized controlled clinical trial (RCT) was to investigate the clinical and biochemical efficacy of a gel containing PDRN and HA used in association with subgingival re-instrumentation in the treatment of residual periodontal pockets.

DETAILED DESCRIPTION:
The aim of the present study was to investigate the clinical and biochemical efficacy of a gel containing polynucleotides (PDRN) and hyaluronic acid (HA) used in association with subgingival re-instrumentation in the treatment of residual periodontal pockets.

50 patients were enrolled in a randomized, split-mouth clinical trial. For each patient, two teeth with similar residual pockets with probing depth (PD) ≥ 5 mm were selected to receive re-instrumentation with (test) or without (control) the adjunctive use of a PDRN and HA based gel. Differences in changes of PD, gingival recession (REC), clinical attachment level (CAL), modified sulcular bleeding index (mSBI), plaque index (PLI) from baseline to 6, 8, 24, 36 and 48 weeks were analyzed and the frequencies of sites with PD <4 mm at 48 weeks were compared. Furthermore, changes in the dosage of alpha-2-macroglobulin (α2M) and of matrix metalloproteinase-9 (MMP-9) from baseline to 6 weeks were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* males and females with ≥ 18 years
* stage 3 generalized periodontitis
* 3-6 months after step 1 and 2 of periodontal treatment, at least two non-adjacent teeth showing one residual pocket with probing depth (PD) ≥5, without mobility and without furcation involvement.

Exclusion Criteria:

* full-mouth plaque score (FMPS) and full-mouth bleeding score (FMBS) >20%
* inadequate restorative therapy or malocclusion
* uncontrolled systemic disease
* immunosuppressive therapy or therapy with corticosteroid or with bisphosphonates
* inflammatory and autoimmune diseases of the oral cavity
* history of malignancy, radiation therapy or chemotherapy for malignancy in the last 5 years
* insulin-dependent diabetes;
* smoking (> 10 cigarettes per day)
* drug and alcohol abuse
* pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2019-09-09 (Actual); Study Completion 2019-12-13 (Actual)

PRIMARY OUTCOMES:
Pocket depth | 12 months
  Clinical evaluations were performed by a blind calibrated examiner, different from the investigator who performed the treatment. At baseline (visit 1) and at 6 (visit 2), 8(visit 3), 24 (visit 4), 36 (visit 5) and 48 (visit 6) weeks using a periodontal probe

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Department of Oral and Maxillofacial Sciences. Section of Periodontics.Sapienza, University of Rome, Rome, Italy